CLINICAL TRIAL: NCT05166876
Title: A Phase II, Randomized, Assessor-blind, Multicenter, Multi-dose, Placebo-controlled Study Assessing the Safety and Anti-coronavirus Response of Brequinar Combined With Dipyridamole in Patients With Mild to Moderate SARS-CoV-2 Infection.
Brief Title: Brequinar Combined With Dipyridamole in Patients With Mild to Moderate COVID-19
Acronym: CCBCRISIS04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low prevalence of COVID-19 in India led to lack of eligible subjects.
Sponsor: Clear Creek Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCB-CRISIS-04
Record Dates: First submitted 2021-12-16; First posted 2021-12-22 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Oral antiviral; DHODH Inhibitor; brequinar
MeSH Terms: conditions — COVID-19 | interventions — brequinar; Dipyridamole

STUDY DESIGN:
Intervention Model Description: All subjects will receive standard of care. In addition, subjects will be randomly assigned to one of 3 treatments: brequinar (50 mg, 100 mg, 150 mg, or 200 mg), placebo (50 mg, 100 mg, 150 mg, or 200 mg), or brequinar + dipyridamole (75 mg TID) in a 2:1:1 ratio in Part 1 of the study using a dose escalation approach. An expansion cohort is planned with the highest safe brequinar dose.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All staff will be blinded to treatment with the exception of the pharmacist and any staff recording study drug administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brequinar monotherapy (Experimental): Brequinar oral capsules will be administered once daily for 5 days using a dose-escalation approach. Planned doses include 50 mg, 100 mg, 150 mg, and 200 mg. Dosing will start at 50 mg and be escalated to the next higher dose if cohort stopping rules are not met.
  Interventions: Drug: Brequinar Sodium
- Placebo (Placebo Comparator): Placebo matching brequinar oral capsules will be administered once daily for 5 days using a dose-escalation approach. Planned doses include 50 mg, 100 mg, 150 mg, and 200 mg. Dosing will start at 50 mg and be escalated to the next higher dose if cohort stopping rules are not met.
  Interventions: Drug: Placebo
- Brequinar-Dipyridamole Combination (Experimental): Brequinar oral capsules will be administered once daily for 5 days using a dose-escalation approach. Planned doses include 50 mg, 100 mg, 150 mg, and 200 mg. Dosing will start at 50 mg and be escalated to the next higher dose if cohort stopping rules are not met. All subjects assigned to this arm will also receive dipyridamole 75 mg tablets TID.
  Interventions: Drug: Brequinar Sodium; Drug: Dipyridamole 75 MG

INTERVENTIONS:
Drug: Brequinar Sodium — 50 mg, 100 mg, 150 mg, 200 mg x 5 days
  Arms: Brequinar monotherapy; Brequinar-Dipyridamole Combination
Drug: Dipyridamole 75 MG — 75 mg TID for 5 days
  Arms: Brequinar-Dipyridamole Combination
Drug: Placebo — 50 mg, 100 mg, 150 mg, 200 mg x 5 days
  Arms: Placebo

SUMMARY:
A Phase 2 multi-center, assessor-blind, randomized study to assess the safety, tolerability, and antiviral activity of brequinar in combination with dipyridamole.

DETAILED DESCRIPTION:
This is a Phase 2 clinical trial in two parts. The first part of the trial will study up to 64 subjects using a dose escalation approach, with 16 subjects per cohort for up to 4 cohorts. The brequinar dose will start at 50 mg per day in Cohort 1, escalating in the next cohort of 16 to 100 mg, then to 150 mg, and finally to 200 mg if safety parameters are met. The dipyridamole dose will be 75 mg three times a day (TID) for subjects assigned to the combination arm for all cohorts. All subjects will also receive standard of care (SOC) for treatment of patients with COVID-19 infection. After identifying the highest brequinar dose that is safe and well tolerated, 48 subjects will be treated in an expansion part comparing the chosen brequinar dose in combination with 75 mg dipyridamole TID to the chosen dose of brequinar alone. The combination of brequinar and dipyridamole shows potent in vitro antiviral activity by blocking DHODH and the pyrimidine salvage pathway, respectively, and the purpose of this study is to establish the safety and antiviral effect of the combination.

During the dose escalation part of the study, subjects with confirmed mild to moderate COVID-19 will receive 5 days of one of the following oral doses: brequinar alone, brequinar in combination with dipyridamole, or placebo. Subjects will have a Screening Visit followed as soon as possible with Study Day 1. Study visits (virtual or in person) will take place at Screening and on specified days. The visits that include bloodwork must be conducted at the study site or arrangements made for sample collection at the subject's home or other appropriate location. Other visits/visit activities for that visit may be conducted remotely using telemedicine or other remote technique. A viral load sample, vital signs (respiratory rate, heart rate, body temperature and SpO2), and a symptom assessment will be completed on specified days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent for the trial, written, electronic, verbal, or other method deemed acceptable by the institution and IRB.
2. Subjects between ≥18 and ≤65 years of age.
3. Subjects found positive for SARS-CoV-2 either by rapid antigen test or by reverse transcription polymerase chain reaction (RT-PCR) using ICMR-validated kit.

   Note: Test need not be repeated in those with possession of confirmed positive report, but positive result test date must be ≤5 days of first dose of study drug.
4. Mild or Moderate COVID-19 as per latest updated version of CLINICAL MANAGEMENT PROTOCOL for COVID-19 (in adults) released by Government of India Ministry of Health and Family Welfare Directorate General of Health Services (EMR Division).
5. The effects of brequinar on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and for 90 days after completion of brequinar administration.
6. Male subjects must agree to refrain from sperm donation and female subjects must agree to refrain from ovum donation from initial study drug administration until 90 days after the last dose of brequinar.
7. At least one non-respiratory COVID-19 symptom characterized as mild to moderate by the Investigator including but not limited to fatigue, chills, fever, body aches, nasal congestion, nausea, vomiting, or other sign or symptom commonly associated with COVID-19 in the opinion of the investigator. Symptom onset must be ≤5 days prior to first dose. Subject must have one or more signs/symptoms present at first dose.
8. Willing to participate in the PK subset if at one of the identified sites.
9. Able to swallow capsules.

Exclusion Criteria:

* 1. Have an oxygen saturation of <90% while breathing ambient air. 2. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject.

  3. Nursing women or women of childbearing potential (WOCBP) with a positive pregnancy test.

  4. Treatment with another DHODH inhibitor (e.g., leflunomide, teriflunomide) or other agents known to cause bone marrow suppression leading to thrombocytopenia.

  5. Ongoing treatment with aspirin and or dipyridamole, famotidine or cimetidine. Remdesivir and ivermectin are prohibited through Study Day 8. Steroids are permitted per the guidelines.

  6. Platelets ≤125,000 cell/mm3. 7. Hemoglobin <10 gm/dL. 8. Absolute neutrophil count <1000 cells/mm3. 9. Renal dysfunction, i.e., creatinine clearance <30 mL/min. 10. AST or ALT >3 x ULN, or total bilirubin >ULN. Gilbert's Syndrome is allowed.

  11. Bleeding disorders or blood loss requiring transfusion in the six weeks preceding enrollment.

  12. Ongoing gastrointestinal ulcer, or gastrointestinal bleeding within 6 weeks of first dose.

  13. Chronic hepatitis B infection, active hepatitis C infection, active liver disease and/or cirrhosis per subject report.

  14. Heart failure, current uncontrolled cardiovascular disease, including unstable angina, uncontrolled arrhythmias, major adverse cardiac event within 6 months (e.g., stroke, myocardial infarction, hospitalization due to heart failure, or revascularization procedure).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - RIMS - Government Medical College, Srikakulam, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Global Hospital, Surat, Gujarat
  - Rajarajeshwari Medical College and Hospital, Bangalore, Karnataka
  - JIPMER Hospital, Puducherry, Puducherry
  - Noble Hospital, Hadapsar, Pune
  - Panimalar Hospital, Chennai, Tamil Nadu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 participants were enrolled at 4 medical clinics in India. First participant was enrolled 02/01/2022, last participant completed the study 06/04/2022.
Period: Overall Study
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Started | 7 | 6 | 13
Completed | 6 | 6 | 13
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination | Total
Number analyzed (Participants) | 7 | 6 | 13 | 26
Age, Continuous [Median (Standard Deviation); unit: years] | 31.00 (14.05) | 53.50 (12.55) | 43.00 (14.12) | 41.00 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 6 | 3 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 6 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 7 | 6 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Brequinar-dipyridamole Combination in COVID-19 Subjects
Description: There were no subjects who experienced grade 3 and 4 toxicities and serious adverse events (SAEs) considered by the investigator to be related to the combination, brequinar alone or placebo alone. therefore frequencies of these events could not be compared.
Time Frame: Day 29
Population: No subjects experienced any grade 3 or 4 toxicity (related adverse event) or serious adverse event (SAE), therefore no analyses could be conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 7 | 6 | 13
Participants | 0 | 0 | 0

2. Secondary Outcome: Reduction of SARS-CoV-2 Levels Using qPCR Through Day 29 and at Days 4, 8, 12, 15, 22, and 29
Description: There were no subjects with detectable viral load after baseline, therefore no analyses could be conducted regarding change in viral load from baseline of SARS-CoV-2 levels using qPCR SARS-CoV-2 levels through Day 29 and at days 4, 8, 12, 15, 22, and 29
Time Frame: Day 29
Population: There were no subjects with detectable viral load after baseline therefore no analyses could be conducted regarding change in viral load.
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Reduction in Time to Symptom Improvement
Description: There were no subjects who had changes in symptom improvement, therefore no analyses of changes in symptom improvement could be conducted.
Time Frame: Day 29
Population: There were no subjects with clinically significant symptoms after baseline therefore no analyses could be conducted regarding change from baseline.
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Reduction in Percentage of Subjects Requiring Hospital Admission/Re-admission as an In-patient for >24 Hours
Description: There were no subjects who required hospital admission/re-admission as an in-patient for >24 hours, therefore no analyses could be conducted for comparative change in percentage of subjects who required hospital admission/readmission for >24 hours.
Time Frame: Day 29
Population: No subjects were hospitalized in any of the groups, therefore no analyses could be conducted.
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Reduction in Percentage of Subjects Requiring Medical Attended Visits, e.g., Hospitalization, Emergency Room Visits, Urgent Care/Family Doctor Visits
Description: There were no subjects requiring medical attended visits, e.g., hospitalization, emergency room visits, Urgent Care/Family Doctor visits, therefore no analyses could be conducted for comparative change in percentage of subjects requiring medical attended visits, e.g., hospitalization, emergency room visits, Urgent Care/Family Doctor visits
Time Frame: Day 29
Population: No subjects required medical attended visits in any of the groups, therefore no analyses could be conducted.
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Reduction in Percentage of Subjects Requiring Supplemental Support Such as Oxygen
Description: There were no subjects that required supplemental support such as oxygen, therefore analyses of comparative change in percentage of subjects requiring supplemental support such as oxygen could not be conducted.
Time Frame: Day 29
Population: No subjects required oxygen in any of the groups, therefore no analyses could be conducted.
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 29 days
Description: Adverse Events (AEs) were collected from the time of first dose of study drug through Day 29. AEs determined by the Investigator to be related to study drug were followed until resolution or until they were considered stable or for at least 30 days after discontinuation of study drug. All AEs recorded on the electronic case report form (eCRF) were coded using the MedDRA dictionary Version 23.1 (or a later version if updated during the study).
Arm/Group | Brequinar Monotherapy | Placebo | Brequinar-Dipyridamole Combination
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 1/7 | 3/6 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brequinar Monotherapy (N=7) | Placebo (N=6) | Brequinar-Dipyridamole Combination (N=13)
Headache (Nervous system disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
Asthenia (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT05166876/Prot_SAP_000.pdf